CLINICAL TRIAL: NCT00722514
Title: Evaluation of a Patient Education Program for Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehazentrum Bad Eilsen (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Dr. Inge Ehlebracht-König, Rehazentrum Bad Eilsen
Other Study IDs: 0110599604
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-07

CONDITIONS: Ankylosing Spondylitis; Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Patient Education as Topic; Standard of Care

ARMS (2):
- IG (Experimental): Patient education
  Interventions: Behavioral: patient education
- CG (Other): without patient education
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: patient education — * complex individual antiinflammatory rehabilitation program during inpatient rehabilitation (physiotherapy, physical therapy, occupational therapy, health-promoting measures and more) and additionally
  * Patient education 6 x 90 Minutes
  Arms: IG
Behavioral: Standard Care — * complex individual antiinflammatory rehabilitation program during inpatient
  * complex individual medical rehabilitation (physiotherapy, physical therapy, occupational therapy, health-promoting measures and more) and additionally
  * further 6 treatments from available disciplines(e.g. massage, electrotherapy, bath)
  Arms: CG

SUMMARY:
Long term disease management is essential for Ankylosing Spondylitis (AS), a chronic progressive systemic inflammatory disease of the axial skeleton. Extensive information about the disease is a necessary first step. An education program for AS was implemented to improve inpatient medical rehabilitation. In a controlled quasi-experimental multicentric study the efficacy of this program was analysed.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing Spondylitis (AS) according to modified New York Criteria
* Early diagnosis criteria for AS
* ESSG Criteria for Spondyloarthritis

Exclusion Criteria:

* History of malignant disease during past five years
* Secondary fibromyalgia syndrome
* Group integration deficiencies
* Seminar repeaters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Primary Completion 2001-02; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Overall Officials: Inge Ehlebracht-Koenig, MD, Principal Investigator — Rehazentrum Bad Eilsen
Locations (1):
- Rehazentrum Bad Eilsen, Bad Eilsen, Lower Saxony, Germany